CLINICAL TRIAL: NCT02829619
Title: Meal Timing, Genetics and Weight Loss in a Mediterranean Population
Brief Title: Meal Timing, Genetics and Weight Loss
Acronym: ONTIME
Status: Recruiting | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, PROF. MARTA GARAULET AZA, Full Professor, Universidad de Murcia
Other Study IDs: R01DK105072-1; R01DK105072 (NIH)
Record Dates: First submitted 2016-06-10; First posted 2016-07-12 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: Obesity; Nutrigenetics; Food Timing; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, saliva
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Meal times differ from culture to culture. These differences may influence energy regulation and, consequently, body weight. Current studies support the notion that not only "what" but also "when" the investigators eat may have a significant role in obesity treatment. Recently, it has been shown that eating the main meal of the day, lunch in Spain, late in the day is predictive of difficulty in weight loss and decreased insulin sensitivity. This project aims to study in a Mediterranean population the potential influence of genetics and food timing on obesity, metabolic syndrome and weight loss.

DETAILED DESCRIPTION:
Meal times differ from culture to culture. These differences may influence energy regulation and, consequently, body weight. Current studies support the notion that not only "what" but also "when" the investigators eat may have a significant role in obesity treatment. Recently, it has been shown that eating the main meal of the day, lunch in Spain, late in the day is predictive of difficulty in weight loss and decreased insulin sensitivity. Furthermore, it has been shown that eating late at night when plasma melatonin concentrations are elevated, impairs glucose tolerance, particularly in MTNR1B risk allele carriers.

The main objective is to identify the mechanisms underlying the association between the timing of food intake, obesity and metabolic syndrome (MetS) in order to design effective weight loss therapies. The long-term goal is to determine the potential impact of more European, i.e., earlier meal timing on obesity, MetS and weight loss.

The challenge for the society is to develop evidence-based dietary interventions incorporating meal timing and genotype to combat the epidemic of obesity and MetS.

These goals will be achieved through three specific approaches:

* Epidemiological (observational study) (Aim 1): To assess in an obese population (n=5000) who will follow a weight loss program if clock-related (CLOCK, PER2, CRY, etc.) and melatonin-related variants (MTNR1B) interact with the timing of food intake to determine weight loss effectiveness and MetS features.
* Interventional (randomized controlled trials) (Aim 2): To determine the internal mechanisms of energy balance and circadian system implicated in the differential effects of food timing (lunch) on weight loss, MetS alterations and the intestinal microbiota (n=25), and to study the potential interaction between meal timing (dinner) and genetic variants MTNR1B for glucose tolerance in obese women (n=100).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: >25 kg/m2
* Age: >18 years of age
* Caucasian

Exclusion Criteria:

* Receiving treatment with thermogenic, lipogenic, or contraceptive drugs
* Diabetes mellitus, chronic renal failure, hepatic diseases, or cancer diagnosis
* bulimia diagnosis, prone to binge eating
* undergoing treatment with anxiolytic or antidepressant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants are voluntarily attending five weight loss clinics in Spain for dietetic and behavioral treatment based upon the principles of a Mediterranean diet . All participants are from the Spanish city of Murcia, located on the Southeast coast of the Mediterranean Sea.
Sampling Method: Probability Sample
Enrollment: 5788 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Total weight loss | weekly, during the 28 weeks of treatment
  Body weight will be measured in barefoot wearing light clothes, with a digital scale to the nearest 0.1 kg, at the same time each day.
Long term weight loss maintenance | once at least one year after ending the treatment
  Body weight will be measured in barefoot wearing light clothes, with a digital scale to the nearest 0.1 kg.

SECONDARY OUTCOMES:
Food timing | at baseline
  Timing of breakfast, lunch and dinner
Sleep timing | at baseline
  Habitual sleep timing is estimated using a self-reported questionnaire.
Siesta timing questionnaire | at baseline
  Habitual siesta timing is estimated using a self-reported questionnaire.
Individual chronotype questionnaire | at baseline
  With the Morning and Eveningness Questionnaire (MEQ)
Food habits questionnaire | at baseline
  Variety of food groups is assessed by at 24h recall the day before starting the intervention and by a a seven days dietary record during the intervention. The number of different food items per day will be counted to assess variety of food
Total energy intake dietary questionnaire | at baseline
  by at 24h recall the day before starting the intervention and by a a seven days dietary record during the intervention. Daily energy intake will be calculated
Macronutrient distribution dietary questionnaire | at baseline
  by at 24h recall the day before starting the intervention and by a a seven days dietary record during the intervention. Macronutrient (% from total calories of the diet) and (grams) will be calculated
Glycemic Index questionnaire | at baseline
  by at 24h recall the day before starting the intervention and by a a seven days dietary record during the intervention. The glycemic index will be calculated by using different composition tables
Barriers to Weight Loss checklist | at baseline
  A questionnaire will be complete by the participants. The test consisted of 29 questions classified into seven sections: meal recording; weight control and weekly interviews; eating habits; portion size; food and drink choice; way of eating; and other obstacles to weight loss. There are were three possible responses (never 0, sometimes 1, very often 2) to those questions that represented barriers to losing weight, such as ''Have you lost your motivation?'' or ''Do you have binges?'' Questions that represented aids to weight loss, such as ''Do you accurately measure your portions?'' or ''Is absolutely everything written down?'' applied the same score (0 to 2) but with negative signs. A final ''Barriers to Weight Loss'' score is calculated by adding every answer's score for each patient.
Emotional eating questionnaire | at baseline
  The EEQ (Emotional eating Questionnaire) will be used extent emotions affect eating behaviour. . All the questions had four possible replies: 1) Never, 2) Sometimes; 3) Generally and 4) Always. Each reply was given a score of 1 to 4, the lower the score, the healthier the behaviour. For the clinical practice subjects are classified in four groups attending to the score obtained. Score between 0-5: non-emotional eater. Score between 6-10: low emotional eater. Score between 11-20: emotional eater. Score between 21-30: very emotional eater.
Physical activity questionnaire | at baseline
  by the IPAQ (international Physical Activity Questionnaire)
Mediterranean Diet Score questionnaire | at baseline
  By the questionnaire developed by Antonia Trichopoulou, M.D., Tina Costacou, Ph.D., Christina Bamia, Ph.D., and Dimitrios Trichopoulos, M.D.
  N Engl J Med 2003; 348:2599-2608June 26, 2003DOI: 10.1056/NEJMoa025039
Glucose tolerance | from 1 year to 3 years after weight loss treatment
  either by meal test or by glucose tolerance test
Daily rhythms of wrist temperature | from 3 months to 3 years after weight loss treatment
  7 day-record of wrist temperature by wrist temperature sensors.
Daily rhythms of activity | from 3 months to 3 years after weight loss treatment
  7 day-record of activity by actiwatch
Daily rhythms of autonomus system by ambulatory electrocardiography | from 3 months to 3 years after weight loss treatment
  7 days of ambulatory electrocardiography
Glucose | at baseline
  Fasting glucose
Insulin | at baseline
  Fasting insulin

CONTACTS AND LOCATIONS:
Overall Officials: Marta Garaulet, PHD, Principal Investigator — Universidad de Murcia
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garaulet M, Vera B, Bonnet-Rubio G, Gomez-Abellan P, Lee YC, Ordovas JM. Lunch eating predicts weight-loss effectiveness in carriers of the common allele at PERILIPIN1: the ONTIME (Obesity, Nutrigenetics, Timing, Mediterranean) study. Am J Clin Nutr. 2016 Oct;104(4):1160-1166. doi: 10.3945/ajcn.116.134528. Epub 2016 Sep 14. PMID 27629052
- [Background] Gomez-Santos C, Saura CB, Lucas JA, Castell P, Madrid JA, Garaulet M. Menopause status is associated with circadian- and sleep-related alterations. Menopause. 2016 Jun;23(6):682-90. doi: 10.1097/GME.0000000000000612. PMID 27093617
- [Background] Corbalan-Tutau MD, Gomez-Abellan P, Madrid JA, Canteras M, Ordovas JM, Garaulet M. Toward a chronobiological characterization of obesity and metabolic syndrome in clinical practice. Clin Nutr. 2015 Jun;34(3):477-83. doi: 10.1016/j.clnu.2014.05.007. Epub 2014 May 28. PMID 24953771
- [Background] Lopez-Guimera G, Dashti HS, Smith CE, Sanchez-Carracedo D, Ordovas JM, Garaulet M. CLOCK 3111 T/C SNP interacts with emotional eating behavior for weight-loss in a Mediterranean population. PLoS One. 2014 Jun 6;9(6):e99152. doi: 10.1371/journal.pone.0099152. eCollection 2014. PMID 24905098
- [Background] Dashti HS, Smith CE, Lee YC, Parnell LD, Lai CQ, Arnett DK, Ordovas JM, Garaulet M. CRY1 circadian gene variant interacts with carbohydrate intake for insulin resistance in two independent populations: Mediterranean and North American. Chronobiol Int. 2014 Jun;31(5):660-7. doi: 10.3109/07420528.2014.886587. Epub 2014 Feb 18. PMID 24548145
- [Background] Bandin C, Martinez-Nicolas A, Ordovas JM, Madrid JA, Garaulet M. Circadian rhythmicity as a predictor of weight-loss effectiveness. Int J Obes (Lond). 2014 Aug;38(8):1083-8. doi: 10.1038/ijo.2013.211. Epub 2013 Nov 15. PMID 24232497
- [Background] Garaulet M, Smith CE, Gomez-Abellan P, Ordovas-Montanes M, Lee YC, Parnell LD, Arnett DK, Ordovas JM. REV-ERB-ALPHA circadian gene variant associates with obesity in two independent populations: Mediterranean and North American. Mol Nutr Food Res. 2014 Apr;58(4):821-9. doi: 10.1002/mnfr.201300361. Epub 2013 Oct 31. PMID 24173768
- [Background] Garaulet M, Gomez-Abellan P. Chronobiology and obesity. Nutr Hosp. 2013 Sep;28 Suppl 5:114-20. doi: 10.3305/nh.2013.28.sup5.6926. PMID 24010751
- [Background] Morales-Falo EM, Sanchez-Moreno C, Esteban A, Alburquerque JJ, Garaulet M. [Quality of the diet "before and during" a weight loss treatment based on Mediterranean Diet; behavioural therapy and nutritional education]. Nutr Hosp. 2013 Jul-Aug;28(4):980-7. doi: 10.3305/nh.2013.28.4.6665. Spanish. PMID 23889612
- [Background] Garaulet M, Gomez-Abellan P, Alburquerque-Bejar JJ, Lee YC, Ordovas JM, Scheer FA. Timing of food intake predicts weight loss effectiveness. Int J Obes (Lond). 2013 Apr;37(4):604-11. doi: 10.1038/ijo.2012.229. Epub 2013 Jan 29. PMID 23357955
- [Background] Bandin C, Martinez-Nicolas A, Ordovas JM, Ros Lucas JA, Castell P, Silvente T, Madrid JA, Garaulet M. Differences in circadian rhythmicity in CLOCK 3111T/C genetic variants in moderate obese women as assessed by thermometry, actimetry and body position. Int J Obes (Lond). 2013 Aug;37(8):1044-50. doi: 10.1038/ijo.2012.180. Epub 2012 Nov 20. PMID 23183326
- [Background] Milagro FI, Gomez-Abellan P, Campion J, Martinez JA, Ordovas JM, Garaulet M. CLOCK, PER2 and BMAL1 DNA methylation: association with obesity and metabolic syndrome characteristics and monounsaturated fat intake. Chronobiol Int. 2012 Nov;29(9):1180-94. doi: 10.3109/07420528.2012.719967. Epub 2012 Sep 24. PMID 23003921
- [Background] Garaulet M, Canteras M, Morales E, Lopez-Guimera G, Sanchez-Carracedo D, Corbalan-Tutau MD. Validation of a questionnaire on emotional eating for use in cases of obesity: the Emotional Eater Questionnaire (EEQ). Nutr Hosp. 2012 Mar-Apr;27(2):645-51. doi: 10.1590/S0212-16112012000200043. PMID 22732995
- [Background] Corbalan-Tutau D, Madrid JA, Nicolas F, Garaulet M. Daily profile in two circadian markers "melatonin and cortisol" and associations with metabolic syndrome components. Physiol Behav. 2014 Jan 17;123:231-5. doi: 10.1016/j.physbeh.2012.06.005. Epub 2012 Jun 15. PMID 22705307
- [Background] Corbalan-Tutau MD, Madrid JA, Garaulet M. Timing and duration of sleep and meals in obese and normal weight women. Association with increase blood pressure. Appetite. 2012 Aug;59(1):9-16. doi: 10.1016/j.appet.2012.03.015. Epub 2012 Mar 23. PMID 22450522
- [Background] Garaulet M, Esteban Tardido A, Lee YC, Smith CE, Parnell LD, Ordovas JM. SIRT1 and CLOCK 3111T> C combined genotype is associated with evening preference and weight loss resistance in a behavioral therapy treatment for obesity. Int J Obes (Lond). 2012 Nov;36(11):1436-41. doi: 10.1038/ijo.2011.270. Epub 2012 Feb 7. PMID 22310473
- [Background] Garaulet M, Smith CE, Hernandez-Gonzalez T, Lee YC, Ordovas JM. PPARgamma Pro12Ala interacts with fat intake for obesity and weight loss in a behavioural treatment based on the Mediterranean diet. Mol Nutr Food Res. 2011 Dec;55(12):1771-9. doi: 10.1002/mnfr.201100437. Epub 2011 Nov 21. PMID 22102511
- [Background] Corbalan-Tutau MD, Madrid JA, Ordovas JM, Smith CE, Nicolas F, Garaulet M. Differences in daily rhythms of wrist temperature between obese and normal-weight women: associations with metabolic syndrome features. Chronobiol Int. 2011 May;28(5):425-33. doi: 10.3109/07420528.2011.574766. PMID 21721858
- [Background] Smith CE, Ordovas JM, Sanchez-Moreno C, Lee YC, Garaulet M. Apolipoprotein A-II polymorphism: relationships to behavioural and hormonal mediators of obesity. Int J Obes (Lond). 2012 Jan;36(1):130-6. doi: 10.1038/ijo.2011.24. Epub 2011 Mar 8. PMID 21386805
- [Background] Sanchez-Moreno C, Ordovas JM, Smith CE, Baraza JC, Lee YC, Garaulet M. APOA5 gene variation interacts with dietary fat intake to modulate obesity and circulating triglycerides in a Mediterranean population. J Nutr. 2011 Mar;141(3):380-5. doi: 10.3945/jn.110.130344. Epub 2011 Jan 5. PMID 21209257
- [Background] Garaulet M, Corbalan-Tutau MD, Madrid JA, Baraza JC, Parnell LD, Lee YC, Ordovas JM. PERIOD2 variants are associated with abdominal obesity, psycho-behavioral factors, and attrition in the dietary treatment of obesity. J Am Diet Assoc. 2010 Jun;110(6):917-21. doi: 10.1016/j.jada.2010.03.017. PMID 20497782
- [Background] Garaulet M, Corbalan MD, Madrid JA, Morales E, Baraza JC, Lee YC, Ordovas JM. CLOCK gene is implicated in weight reduction in obese patients participating in a dietary programme based on the Mediterranean diet. Int J Obes (Lond). 2010 Mar;34(3):516-23. doi: 10.1038/ijo.2009.255. Epub 2010 Jan 12. PMID 20065968
- [Background] Garaulet M, Lee YC, Shen J, Parnell LD, Arnett DK, Tsai MY, Lai CQ, Ordovas JM. CLOCK genetic variation and metabolic syndrome risk: modulation by monounsaturated fatty acids. Am J Clin Nutr. 2009 Dec;90(6):1466-75. doi: 10.3945/ajcn.2009.27536. Epub 2009 Oct 21. PMID 19846548
- [Background] Gomez-Abellan P, Hernandez-Morante JJ, Lujan JA, Madrid JA, Garaulet M. Clock genes are implicated in the human metabolic syndrome. Int J Obes (Lond). 2008 Jan;32(1):121-8. doi: 10.1038/sj.ijo.0803689. Epub 2007 Jul 24. PMID 17653067
- [Background] Lo MT, Bandin C, Yang HW, Scheer FAJL, Hu K, Garaulet M. CLOCK 3111T/C genetic variant influences the daily rhythm of autonomic nervous function: relevance to body weight control. Int J Obes (Lond). 2018 Feb;42(2):190-197. doi: 10.1038/ijo.2017.168. Epub 2017 Jul 24. PMID 28736443
- [Background] Bonnet G, Gomez-Abellan P, Vera B, Sanchez-Romera JF, Hernandez-Martinez AM, Sookoian S, Pirola CJ, Garaulet M. Serotonin-transporter promoter polymorphism modulates the ability to control food intake: Effect on total weight loss. Mol Nutr Food Res. 2017 Nov;61(11). doi: 10.1002/mnfr.201700494. Epub 2017 Sep 1. PMID 28766852
- [Background] Vera B, Dashti HS, Gomez-Abellan P, Hernandez-Martinez AM, Esteban A, Scheer FAJL, Saxena R, Garaulet M. Modifiable lifestyle behaviors, but not a genetic risk score, associate with metabolic syndrome in evening chronotypes. Sci Rep. 2018 Jan 17;8(1):945. doi: 10.1038/s41598-017-18268-z. PMID 29343740
- [Background] Dashti HS, Gomez-Abellan P, Qian J, Esteban A, Morales E, Scheer FAJL, Garaulet M. Late eating is associated with cardiometabolic risk traits, obesogenic behaviors, and impaired weight loss. Am J Clin Nutr. 2021 Jan 4;113(1):154-161. doi: 10.1093/ajcn/nqaa264. PMID 33022698
- [Background] Garaulet M, Vizmanos B, Muela T, Betancourt-Nunez A, Bonmati-Carrion MA, Vetter C, Dashti HS, Saxena R, Scheer FAJL. Evening types as determined by subjective and objective measures are more emotional eaters. Obesity (Silver Spring). 2023 May;31(5):1192-1203. doi: 10.1002/oby.23749. PMID 37140408
- [Background] Vizmanos B, Cascales AI, Rodriguez-Martin M, Salmeron D, Morales E, Aragon-Alonso A, Scheer FAJL, Garaulet M. Lifestyle mediators of associations among siestas, obesity, and metabolic health. Obesity (Silver Spring). 2023 May;31(5):1227-1239. doi: 10.1002/oby.23765. PMID 37140401
- [Derived] De la Pena-Armada R, Longo-Silva G, Rodriguez-Martin M, Yang HW, Garaulet M. Key Determinants of Weight Loss Trajectory Across Different Periods of a Behavioral Weight Loss Intervention. Obesity (Silver Spring). 2026 Jan 20. doi: 10.1002/oby.70113. Online ahead of print. PMID 41559528
- [Derived] Rodriguez-Martin M, Szczerbinski L, Garaulet M, Dashti HS. The Effect of Habitual Sleep Duration on Weight Loss during a Behavioral Weight Loss Intervention in a Mediterranean Population. J Nutr. 2025 Nov;155(11):4060-4064. doi: 10.1016/j.tjnut.2025.09.010. Epub 2025 Sep 19. PMID 40976481
- [Derived] Yang HW, De la Pena-Armada R, Sun H, Peng YQ, Lo MT, Scheer FAJL, Hu K, Garaulet M. Uncovering key factors in weight loss effectiveness through machine learning. Int J Obes (Lond). 2025 Jun;49(6):1189-1199. doi: 10.1038/s41366-025-01766-w. Epub 2025 May 6. PMID 40328924
- [Derived] Dashti HS, Scheer FAJL, Saxena R, Garaulet M. Impact of polygenic score for BMI on weight loss effectiveness and genome-wide association analysis. Int J Obes (Lond). 2024 May;48(5):694-701. doi: 10.1038/s41366-024-01470-1. Epub 2024 Jan 24. PMID 38267484